CLINICAL TRIAL: NCT06781255
Title: Evaluation of K9 in Subjects With Diabetic Macular Edema (DME)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michelle Abou-Jaoude (Other)
Collaborators: Inflammasome Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Michelle Abou-Jaoude, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100315
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Kamuvudine-9

STUDY DESIGN:
Masking Description: Unmasked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with DME (Experimental): Patients will receive a regimen of 96 mg tablets of K9 to be taken twice a day for 24 weeks.
  Interventions: Drug: Kamuvudine-9

INTERVENTIONS:
Drug: Kamuvudine-9 — 96 mg tablets taken twice a day for 24 weeks

SUMMARY:
A non-randomized study evaluating the safety of an orally administered inflammasome inhibitor, K9, for the treatment of diabetic macular edema (DME).

DETAILED DESCRIPTION:
This is an twenty-eight (28) week non-randomized, open-label, safety study evaluating twice daily, oral K9 in five (5) patients. Subjects with DME meeting inclusion/exclusion criteria will be offered enrollment into this study. A screening visit and subject selection criteria will be used to assess subject eligibility prior to enrollment. Patients will be supplied with tablets of K9 to be taken orally BID for 24 weeks. Safety will be assessed over a series of visits over an 28 week period.

ELIGIBILITY:
Inclusion Criteria:

* BCVA of ≥ 24 and ≤ 73 letters (20/40 or worse but at least 20/320) by an ETDRS chart. BCVA of the non-study eye must be no worse than 20/400 Snellen equivalent)
* Diagnosis of diabetes mellitus, type 1 or 2 with non-proliferative or non-high risk proliferative diabetic retinopathy. Any one of the following will be considered sufficient evidence that diabetes is present:
* Current regular use of insulin for the treatment of diabetes
* Current regular use of oral hypoglycemic agents for the treatment of diabetes
* DME based on investigator's clinical evaluation and demonstrated on fundus photographs, fluorescein angiograms, and/or spectral domain-optical coherence tomography (SD-OCT)
* Mean foveal thickness of at least 325 µm by SD-OCT
* Ability and willingness to comply with the treatment and follow up procedures
* Ability to understand and sign the informed consent form
* Intraocular pressure of ≤ 21 mm Hg on 2 or fewer IOP lowering medications

Exclusion Criteria:

* Pregnant patients, currently lactating patients, or females of childbearing potential (unless using reliable contraception such as double barrier, surgical sterilization, oral contraceptives, intrauterine device (IUD), etc.
* Body weight less than 55 kg
* Allergy or hypersensitivity (known or suspected) to fluorescein or any component of the investigational product or delivery system
* Any ocular surgery in the study eye within 12 weeks of screening
* History of vitrectomy in the study eye
* Aphakia in the study eye
* Presence of severe foveal ischemia, defined as foveal avascular zone (FAZ) of >1.5 mm2 on OCT-Angiography
* Prior intraocular or periocular treatment for DME including any of the following:
* Intravitreous injection of anti-VEGF therapies including but not limited to bevacizumab, ranibizumab, aflibercept, faricimab, and/or brolucizumab within the last 1 month
* Intravitreous or sub-Tenon delivery of any steroid therapy (such as triamcinolone, dexamethasone) in the last 6 months or a fluocinolone acetonide implant for 3 years.
* Macular laser for the treatment of diabetic macular edema within 6 months of screening
* Any change in systemic steroidal therapy within 3 months of screening
* Retinal or choroidal neovascularization due to ocular conditions other than diabetic retinopathy (e.g. presumed ocular histoplasmosis, high myopia (spherical equivalent greater than 8 diopters), macular degeneration)
* History or presence of viral disease of the cornea or conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, any mycobacterial infections of the eye, or any fungal disease of any ocular structure or history of infectious retinitis
* History or presence of any disease or condition that in the investigator's opinion would preclude study treatment or follow-up or that in the opinion of the investigator would render them as unlikely to benefit from study treatment.
* History or presence of any other condition except for DME that could affect interpretation of study assessments (for example, but not limited to, geographic atrophy, macular hole, macular pucker, foveomacular traction, retinal vein occlusion, retinal degenerations)
* Any lens or corneal opacity which impairs visualization of the posterior pole
* Participation in another clinical trial within 12 weeks before the screening visit or during the study
* History of any clinically significant medical disorders the principal investigator considers exclusionary, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, neoplastic disease, renal or urinary tract diseases, or dermatological disease.
* History or current evidence of hypersensitivity to any components of the study medication, as assessed by the investigator.
* Participation in any systemic experimental treatment or any other systemic investigational new drug within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
* Expectation that subject will be moving away from the area of the clinical treatment center without the ability to return for visits within the study period

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 28 weeks
  Frequency of participants experiencing ocular or systemic adverse events.
Change from baseline in central subfield thickness (CST) | Screening (baseline), Day 1 Visit, and weeks 6, 12, 18, and 24
  Central subfield thickness (CST) measured on spectral domain-optical coherence tomography (SD-OCT)
Mean change from baseline in best corrected visual acuity (BCVA) | Screening (baseline), Day 1 Visit, and weeks 6, 12, 18, and 24
  Mean change from baseline assessed by the ETDRS chart. Best-corrected visual acuity as defined by the number of letters read on the scale set by the ETDRS (Early Treatment of Diabetic Retinopathy Study). (More letters read equates to better visual acuity)

SECONDARY OUTCOMES:
Change from baseline in macular volume on spectral domain-optical coherence tomography (SD-OCT) | Screening (baseline), Day 1 Visit, and weeks 6, 12, 18, and 24
  This equipment is used to take photos of the retina layer of the eye and provides two- and three-dimensional images by using near-infrared, broad-bandwidth light source to illuminate the retina. This will be used to look for mean changes from baseline for a change in conditions in eyesight.
Change from baseline in retinal thickening on fundus photography | Screening (baseline), and weeks 6, 12, 18, and 24
  This equipment is used to take high-resolution, ultra-wide field images of the retina to look at the entirety of the back of the eye. This will be used to look for mean changes from baseline for a change in conditions in eyesight
Change from baseline in hard exudates in lesion involving the macula on fundus photography | Screening (baseline), and weeks 6, 12, 18, and 24
  This equipment is used to take high-resolution, ultra-wide field images of the retina to look at the entirety of the back of the eye. This will be used to look for mean changes from baseline for a change in conditions in eyesight
Change from baseline in foveal avascular zone on optical coherence tomography angiography (OCT-A) | Screening (baseline), and weeks 6, 12, 18, and 24
  This equipment is used to take photos of multiple layers of the back of your eye and depicts blood vessels and other structures to help the study doctor measure changes from the baseline in your eyesight.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Abou-Jaoude, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No